CLINICAL TRIAL: NCT00170885
Title: Multicenter, Randomized, Open-label Trial to Evaluate the Safety, Tolerability and Efficacy of Two Regimens of Everolimus Plus Cyclosporine Microemulsion, Given According to Different Blood Target Levels, in de Novo Renal Transplant Recipients
Brief Title: Everolimus in Combination With Cyclosporine Microemulsion in de Novo Renal Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis Pharmaceticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AIT02
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation
Keywords: acute rejection; renal function; everolimus; cyclosporine microemulsion
MeSH Terms: interventions — Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
The purpose of the study in de novo renal transplant patients is to evaluate the effect on renal function of an optimized new regimen in comparison with the standard everolimus exposure plus a low-dose cyclosporine microemulsion regimen.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of deceased, living unrelated, or non-human leukocyte antigen (HLA) identical living related donor renal transplant who actually have a viable kidney transplant at the time of randomization (within 24 hours of graft reperfusion)
* The renal cold ischemic time must be < 36 hours.
* The age of the donor must be between 15 and 65 years.

Exclusion Criteria:

* Patients who are recipients of multiple organ transplants, including more than one kidney
* Patients who have previously received an organ transplant which failed within one year
* Patients with current panel reactive T-cell antibody titers of 50% or more
* Patients who are recipients of A-B-O incompatible transplants or T-cell crossmatch positive transplant

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Renal function assessed by glomerular filtration rate before and during the first 6 months of treatment

SECONDARY OUTCOMES:
Pharmacokinetics (PK)
Count of CD4 and CD8 positive lymphocytes
Metabolic control: lipids, glycaemic control, proteinuria, enzymes
Ultrasound ejection fraction
Major adverse cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland

REFERENCES:
- [Result] Ponticelli C, Salvadori M, Scolari MP, Citterio F, Rigotti P, Veneziano A, Bartezaghi M; EVEREST Study. Everolimus and minimization of cyclosporine in renal transplantation: 24-month follow-up of the EVEREST study. Transplantation. 2011 May 27;91(10):e72-3. doi: 10.1097/TP.0b013e318216c1db. No abstract available. PMID 21540717